CLINICAL TRIAL: NCT04126889
Title: Awareness and Knowledge of the Surgical Safety Checklist Among Operational Staff in University Teaching Hospital, Kathmandu, Nepal: A Cross-sectional Questionnaire
Status: Completed | Type: Observational
Sponsor: Fukushima Medical University (Other)
Responsible Party: Principal Investigator, Yurie Kobashi, Principal Investigator, Fukushima Medical University
Other Study IDs: FukushimaMU
Record Dates: First submitted 2019-10-10; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Surgical Checklist
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire survey — questionnaire survey

SUMMARY:
The introduction of the World Health Organization Surgical Safety Checklist (WHO SSC) is a priority to promote surgical safety. However, little is known regarding awareness and knowledge of the WHO SSC in developing countries. This study aimed to obtain region-specific information for the introduction of the checklist in a core medical institution in Nepal.

The present research was a cross-sectional study using data from a survey conducted at the Tribhuvan University Teaching Hospital (TUTH) in Kathmandu, Nepal. A questionnaire was distributed to 150 healthcare professionals working in the operating theatre. Responses to the questionnaire were analysed descriptively and regression analyses identified factors associated with awareness of the checklist.

ELIGIBILITY:
Inclusion Criteria:

* have optimal experience

Exclusion Criteria:

* less experience

Ages: 24 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: health professionals in operation room
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Awareness of Surgical Safety Checklist | 24 weeks
  Whether medical staffs know about Surgical Safety Checklist, Participants can answer to the question for yes or no.

CONTACTS AND LOCATIONS:
Locations (1):
- Tribhuvan University Teaching Hospital, Kathmandu, Nepal